CLINICAL TRIAL: NCT06908486
Title: Assessing Cognitive Bias Modification for Interpretation (CBM-I) on Pain Severity and Interference in People With Type 2 Diabetes and Persistent Pain
Brief Title: Cognitive Bias Modification for Interpretation (CBM-I) in People With Type 2 Diabetes and Persistent Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024/HE000161
Record Dates: First submitted 2025-04-01; First posted 2025-04-03 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes; Persistent Pain
Keywords: cognitive bias modification; interpretation bias; type 2 diabetes; pain
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Bias Modification for Interpretation (Experimental): The Ambiguous Scenarios paradigm is administered remotely online. The intervention is administered four times: at day 1, day 4, day 7, and day 14. Each intervention presents 30 ambiguous scenarios and associated comprehension questions, and should take approximately 20 minutes to complete. All scenarios in this arm are resolved to be benign.
  Interventions: Behavioral: Cognitive Bias Modification for Interpretation
- Placebo Cognitive Bias Modification for Interpretation (Placebo Comparator): The placebo Ambiguous Scenarios paradigm is administered remotely online. The intervention is administered four times: at day 1, day 4, day 7, and day 14. Each intervention presents 30 ambiguous scenarios and associated comprehension questions, and should take approximately 20 minutes to complete. Scenarios are resolved as either benign or pain-related, with equal numbers (15) of each per session.
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Cognitive Bias Modification for Interpretation — Cognitive Bias Modification involves administering the Ambiguous Scenarios paradigm. This is a series of ambiguous scenarios which could be resolved to be associated with pain. The task consists of 30 unique scenarios and an associated comprehension question (pertaining to the pain-relatedness of the scenario), which are presented in a random order to participants.
  Each scenario presents an ambiguous sentence, ending with a word fragment which the participant must complete. The statement remains ambiguous until the completion of the word fragment, which resolves the statement as either pain-related or benign. For example, the statement "You are bush walking. Suddenly, you trip over and fall onto your knees. Your knees feel all wet, and you look down to see..." can be followed by "le_v_s [leaves]" for a benign resolution, or "bl__d [blood]" for a pain-related resolution. In the intervention group, all 30 scenarios will be followed with the benign word fragment.
  Arms: Cognitive Bias Modification for Interpretation
Behavioral: Placebo — The Ambiguous Scenarios paradigm described previously will be used for the placebo intervention. The same 30 scenarios will be presented to participants, however 50% (15) trials will be followed by the benign word fragment, ad 50% (15) trials will be followed by the pain-related word fragment.
  Arms: Placebo Cognitive Bias Modification for Interpretation

SUMMARY:
The goal of this clinical trial is to examine the efficacy of cognitive bias modification for interpretation (CBM-I) in people with Type 2 Diabetes and persistent pain. The main question[s] it aims to answer is whether interpretation bias training away from pain improves pain outcomes.

Participants in the CBM-I group will complete 4 online training sessions approximately half an hour each. Each session will present participants with ambiguous scenarios which may be pain-related, however the final word of the sentence will resolve the scenario as benign (thus training participants to make benign interpretations). A measure of interpretation bias will be administered following the fourth training session, and pain severity and interference will be measured at baseline, post-training, two week follow up, and three month follow up.

The study hypothesises that participants in the CBM-I group will demonstrate a greater reduction in the co-primary outcomes of pain severity and pain interference over time compared to those in the placebo control.

DETAILED DESCRIPTION:
Pre-intervention stage The study will employ a dual consent process. First, participants will complete an "expression of interest" survey which contains the eligibility survey. Given it is crucial for the study to include people with diabetes and persistent pain, this eligibility survey will be used to ensure the sample meets our eligibility criteria of being 1) are over 18 years of age; 2) have been diagnosed with type 2 diabetes; 3) have persistent pain; 4) score ≥ 3 on pain severity subscale on BPI; 5) fluent in English; 6) have access to internet and ability to use a computer over three months.

Participants deemed eligible for the study will be provided with the Participant Information Statement and consent form via Qualtrics, which will provide detailed information about the study, the nature of their participation, and their rights as participants, including the right to withdraw at any point. Participants who do not consent to participate will be redirected to the end-of-survey.

After providing consent, participants will be asked to complete the baseline questionnaires: Brief Pain Inventory (BPI), Depression, Anxiety and Stress Scale (DASS-21), 12-Item Short Form Survey (SF-12), the Worries about Recurrence or Progression Scale (WARPS) and the Treatment adherence perception (TAPQ). The rationale of these measures is that they are theoretically related to interpretation biases and are hypothesised to change following training. This is expected to take approximately 15-20 minutes of their time.

Intervention stage Immediately following completion of baseline questionaries, participants will be randomised to either the CBM-I or placebo groups automatically using a computer algorithm in Qualtrics and invited to participate in the first session (training session 1) (day 1). Neither the participants nor the researchers will be aware of which group the participant has been allocated to.

Three days after completion of the first training session (day 4), participants will be invited via email automated by Qualtrics to the next training session (training session 2). On day 7, participants will be invited to the next training session (training session 3). Each training session is expected to take 10-15 minutes.

On day 14, participants will be invited to the final training session (training session 4), which will be followed immediately by the follow-up questions (follow-up 1). Participants will therefore complete four training sessions in total over the course of 14 days.

Participants will complete the BPI questionnaire prior to each CBM-I training session. Such that, BPI is measured at baseline, prior to CBM-I training session, and at two follow-up points: 2 weeks and 3 months post-intervention.

Note that participants will be asked to complete the training within two days of being email the link. The training sessions are not mandatory, and whether the participants complete each training session they will be still sent the links for the remaining training sessions.

Post-treatment On day 14, following the final training, participants will complete a series of questionnaires: BPI, DASS-21, SF-12, WARPS, TAPQ, Ambiguous cues task, Recognition Task, Post-Intervention Questionnaire. This survey is estimated to take up to approximately 30-35 minutes (inclusive of training time).

Follow-up 1 Exactly two weeks after post-treatment (day 28), participants will be invited via email and asked to complete the follow-up questionnaires (same as baseline), and the post-intervention questionnaire. This is estimated to take 15-20 minutes.

Follow-up 2 Three months after post-treatment, participants will be invited via email and asked to complete the follow-up questionnaires (same as baseline) and the post-intervention questionnaire. This is estimated to take 15-20 minutes. As outlined in the debrief statement, if the CBM-I intervention appears to be beneficial at the conclusion of the study, access to the training will be provided for all placebo group participants.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Have a diagnosis of Type 2 diabetes.
* Have persistent pain (pain present on more days than not, for 3 months or longer).
* Score ≥ 3 on average pain severity on the Brief Pain Inventory (BPI).
* Fluent in English
* Have access to internet and ability to use a computer over a three month period.

Exclusion Criteria:

* Under 18 years of age
* No diagnosis of Type 2 diabetes
* No persistent pain
* Not fluent in English
* No access to internet nor ability to use a computer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Pain severity | Baseline, post intervention (day 14), Pre intervention session 2 (day 4), pre intervention session 3 (day 7) [primary timepoint], two week follow up post intervention (day 28) [primary timepoint], three month post intervention follow up (3 months)
  Intensity subscale of the Brief Pain Inventory (range 0 - 40; lower scores represent less pain severity, i.e. better outcome)
Pain interference | Baseline, post intervention (day 14), Pre intervention session 2 (day 4), pre intervention session 3 (day 7) [primary timepoint], two week follow up post intervention (day 28) [primary timepoint], three month post intervention follow up (3 months)
  Interference subscale of the Brief Pain Inventory (range 0 - 70; lower scores represent less pain interference, i.e. better outcome)

SECONDARY OUTCOMES:
Interpretation bias to pain (1) | Post intervention (day 14)
  Bias score on the Interpretation Bias Recognition Task (range -4 to 4; lower scores represent smaller interpretation bias to pain, i.e. better outcome)
Interpretation bias to pain (2) | Post intervention (day 14)
  Bias score on the Ambiguous Cues task (range from 0 - 14; lower scores represent smaller interpretation bias to pain, i.e. better outcome)
Health-related quality of life | Baseline, post intervention (day 14), 2 week follow up (day 28), 3 month follow up (day 104)
  12 Item Short Form Health Survey score (scores are reported as Z scores, with a mean of 50 and a standard deviation of 10. Scores greater than 50 are indicative of better than average health-related quality of life).
Depression | Baseline, post intervention (day 14), 2 week follow up (day 28), 3 month follow up (day 104)
  Depression subscale of the 21 item Depression Anxiety Stress Scales (range 0 - 21; lower scores represent less depression, i.e. better outcome)
Anxiety | Baseline, post intervention (day 14), 2 week follow up (day 28), 3 month follow up (day 104)
  Anxiety subscale of the 21 item Depression Anxiety Stress Scales (range 0 - 21; lower scores represent less anxiety, i.e. improved outcome)
Stress | Baseline, post intervention (day 14), 2 week follow up (day 28), 3 month follow up (day 104)
  Stress subscale of the 21 item Depression Anxiety Stress Scales (range 0 - 21; lower scores represent less stress, i.e. improved outcome)
Fear of disease progression | Baseline, post intervention (day 14), 2 week follow up (day 28), 3 month follow up (day 104)
  Worries about Recurrence or Progression Scale score (range 18 - 90; lower scores represent less worry about progression, i.e. better outcome)
Treatment Adherence | Baseline, post intervention (day 14), 2 week follow up (day 28), 3 month follow up (day 104)
  Treatment Adherence Perception Questionnaire (range 16 - 97; higher scores represent greater treatment adherence, i.e. better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Louise Sharpe, Principal Investigator — University of Sydney
Locations (1):
- University of Sydney, Camperdown, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification will be made available.
Time Frame: Data will be available immediately following publication, with no determined end date.
Access Criteria: Data will be made available to researchers who specifically request the data, by contacting the authors.